CLINICAL TRIAL: NCT07205510
Title: Sarcopenia, Metabolic Diseases, and Integrated Aging Longitudinal Evaluation (SMILE)
Status: Recruiting | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LY2025-239-A
Record Dates: First submitted 2025-08-28; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Sarcopenia; Metabolic Diseases; All-cause Mortality; Aging; Cardiometabolic Diseases
Keywords: Sarcopenia; Metabolic Diseases; Aging; All-cause mortality; Cardiometabolic Diseases
MeSH Terms: conditions — Sarcopenia; Metabolic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Serum, whole blood, urine, and fecal specimens
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: nothing — This is an observational study.

SUMMARY:
This study aims to establish an ambispective cohort platform centered on the pathological axis of "sarcopenia-metabolic disorders-aging progression", integrating multimodal data including demographic characteristics, lifestyle factors, clinical phenotypes, laboratory tests, medical imaging, and biospecimens. Namely 'Sarcopenia, Metabolic Diseases, and Integrated Aging Longitudinal Evaluation (SMILE)'.

DETAILED DESCRIPTION:
Sarcopenia is an age-related syndrome characterized by progressive decline in skeletal muscle mass, strength, and function. Traditionally regarded as a consequence of aging, it not only impairs physical mobility, nutritional status, and activities of daily living but also significantly increases the risk of falls, frailty, disability, and subsequent hospitalization. Furthermore, sarcopenia is associated with prolonged hospital stays, elevated postoperative complications, and even premature mortality, imposing substantial economic and healthcare burdens on patients, families, and society.

Recent studies have revealed a complex interplay between sarcopenia and metabolic disorders (e.g., diabetes, dyslipidemia, and obesity), which collectively accelerate the aging process and elevate the risks of cardiovascular events, cardiovascular mortality, and all-cause mortality. Therefore, early identification of changes in muscle mass and function, along with preventive measures against sarcopenia, is crucial for mitigating long-term disease risks. However, strategies for early detection of muscle aging progression and at-risk populations remain to be further elucidated.

This study aims to establish an ambispective cohort platform centered on the pathological axis of "sarcopenia-metabolic disorders-aging progression", integrating multimodal data including demographic characteristics, lifestyle factors, clinical phenotypes, laboratory tests, medical imaging, and biospecimens. Namely 'Sarcopenia, Metabolic Diseases, and Integrated Aging Longitudinal Evaluation (SMILE)'. By combining retrospective and prospective cohort analyses, we will longitudinally track individual health data and conduct in-depth exploration of interaction mechanisms. The objectives are to unravel the dynamic interplay between sarcopenia and metabolic diseases in aging. Assess their mid-to-long-term impact on cardiovascular events and all-cause mortality, and develop novel strategies for early identification and risk stratification.

The findings will provide a robust theoretical foundation and key technological support for precision interventions in sarcopenia, delaying functional decline, and optimizing health management in aging populations. This study holds significant implications for addressing chronic disease risks exacerbated by population aging and alleviating associated socioeconomic burdens.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 18 and over

Exclusion Criteria:

1. Does not cooperate in signing the informed consent form;
2. Does not possess legal capacity;
3. In a state of loss of consciousness;
4. Suffering from severe mental illness, unable to communicate normally;
5. The researcher believes that the subject has a disease that affects the assessment of results and is unsuitable for inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients visiting the Geriatrics Department of Renji Hospital affiliated with Shanghai Jiao Tong University School of Medicine, who were aged 18 years and above.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2040-12-31 (Estimated); Study Completion 2040-12-31 (Estimated)

PRIMARY OUTCOMES:
all-cause mortality | From enrollment to the 5-year and 10-year follow-up visit.
  Collect information on all-cause mortality of patients through hospital medical records, telephone follow-ups, outpatient follow-ups, etc., in order to assess the combined effects and underlying mechanisms of sarcopenia, metabolic diseases, and aging on all-cause mortality.

SECONDARY OUTCOMES:
cause-specific mortality | At 5 and 10 years from the baseline visit.
  Collect information on cause-specific mortality of patients through hospital medical records, telephone follow-ups, outpatient follow-ups, etc., in order to assess the combined effects and underlying mechanisms of sarcopenia, metabolic diseases, and aging on cause-specific mortality. In-depth exploration of the role of sarcopenia, metabolic diseases, and aging in the severe outcomes of mortality caused by various diseases.
Major adverse cardiovascular events | At 5 and 10 years from the baseline visit.
  Through medical records within the hospital, telephone follow-ups, outpatient follow-ups, we will collect detailed information on the occurrence of new major adverse cardiovascular events (cardiovascular death, myocardial infarction, stroke) in the study subjects during the follow-up period. The aim is to analyze the impact, mechanisms, and interactions of sarcopenia, metabolic diseases, and aging on the occurrence and development of these adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Geriatrics, Renji Hospital, School of Medicine, Shanghai Jiaotong University, Shanghai, China., Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
Applicants must submit a specific research plan to the research initiator and apply to share the data thereafter.
Supporting Information: Study Protocol, SAP, CSR